CLINICAL TRIAL: NCT07105865
Title: The Role of NIchel and LTPs Sensitization in Functional Gastrointestinal Disorders: the NILT Study
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, MD,PhD,Prof, Federico II University
Other Study IDs: 283/2025
Record Dates: First submitted 2025-07-16; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Food Allergy in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-specific lipid transfer proteins (nsLTPs) are currently recognized as the most prevalent cause of primary IgE-mediated food allergy in Mediterranean populations and constitute a leading trigger of anaphylactic reactions. In Italy, the prevalence of LTP sensitization is estimated at 2-2.4% in adults and approximately 9% in children, with marked geographic variation. Specifically, higher prevalence rates are observed in central and southern regions and on the islands (21.3%-27.2%) compared to the northern regions (approximately 11%).

LTPs are ubiquitous panallergens, widely expressed throughout the plant kingdom. They represent the major allergens within the Rosaceae family in individuals not sensitized to birch pollen and have also been identified and characterized in numerous plant-derived foods, including nuts, legumes, rice, maize, beer, spelt, and wheat. The clinical spectrum of LTP hypersensitivity is highly heterogeneous. While a significant proportion of sensitized individuals remain asymptomatic, others may present with localized reactions such as contact urticaria or oral allergy syndrome (OAS). More severe cases may involve gastrointestinal symptoms (e.g., vomiting, epigastric discomfort, abdominal pain), cutaneous and respiratory manifestations, and systemic responses up to anaphylactic shock.

Nickel is a ubiquitous metal employed in a wide range of industrial applications and consumer products, including stainless steel, metal plating, various alloys, and inexpensive jewelry. It is also naturally present in both animal and plant-based food sources (e.g., cereals, cocoa, legumes, fresh fruits and nuts, fish). Nickel is the most common sensitizer in allergic contact dermatitis, affecting approximately 20% of the general population and around 10% of the pediatric population. Sensitization to nickel involves a delayed-type (Type IV) hypersensitivity reaction and is not IgE-mediated. Clinical manifestations range from localized allergic contact dermatitis to systemic involvement, referred to as systemic nickel allergy syndrome (SNAS), which is characterized predominantly by gastrointestinal symptoms, although respiratory and other systemic manifestations can also occur.

Gastrointestinal symptoms such as gastroesophageal reflux disease (GERD), functional dyspepsia, abdominal pain, and altered bowel habits, when not associated with overt allergic signs or underlying organic disease, are typically classified as functional gastrointestinal disorders (FGIDs). Several studies report that up to 40% of adult patients with FGIDs exhibit nickel sensitization; however, data in the pediatric population remain scarce.

Chelanik® is a dietary supplement designed to support individuals with nickel hypersensitivity. It contains bioactive components purported to exert immunomodulatory and anti-inflammatory effects. Nevertheless, in vitro human data directly demonstrating its activity on lymphocyte function are currently lacking.

This prospective, experimental, single-center study aims to determine the prevalence of sensitization to LTP and nickel among patients presenting with functional dyspepsia or irritable bowel syndrome (IBS), and to assess in vitro the potential immunomodulatory effects of Chelanik® on peripheral blood lymphocytes from individuals with nickel allergy.

ELIGIBILITY:
Inclusion Criteria:

* Age at least of 4 years
* both sexes
* history of functional dyspepsia (according to the Rome IV criteria, at least one symptom among the following - duration of symptoms greater than 4 days per month and for more than 2 consecutive months, feeling of post-prandial fullness, early satiety, pain and/or epigastric burning not associated with defecation - in the absence of organic disease) and irritable bowel syndrome (according to the Rome IV criteria, including all of the following criteria for at least 2 months prior to diagnosis - abdominal pain for at least 4 days per month associated with one/more of the following: change in EF, change in stool shape/appearance, if constipation is noticed, pain does not resolve with resolution of constipation - in the absence of organic disease).
* written informed consent from the parents of the participants and the participants if over 6 years of age.

Exclusion Criteria:

* Age < 4 years
* Evidence of gastrointestinal pathology of organic nature (GERD, Helicobacter Pylori infection, eosinophilic diseases, celiac disease, chronic inflammatory bowel disease, chronic pancreatitis, cholelithiasis, neoplasia); motility disorder on a post-infectious basis; food intolerances (e.g. lactose), carbohydrate malabsorption, use of ASAs, NSAIDs; chronic systemic diseases (diabetes, amyloidosis, neuropathy) and autoimmune diseases; neuropsychiatric disorders; pregnancy.

Ages: 4 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 50 adults (>18 years) and 50 pediatric (4-17 years), of both sexes, belonging to the Adult Gastroenterology Programs and Pediatrics Section of Department of Translational Medical Sciences (University of Naples Federico II).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of nickel and LTP sensitization in patients with symptoms of functional dyspepsia and irritable bowel syndrome | At baseline
  To evaluate the prevalence of nickel and LTP sensitization in patients with symptoms of functional dyspepsia (according to the Rome IV criteria, at least one symptom among the following for at least 4 days at the month and for at least 2 months before diagnosis - feeling of post-prandial fullness, satiety early epigastralgia or heartburn unrelated to defecation - in the absence of organic disease) and irritable bowel syndrome (according to Rome IV criteria, including all of the following for at least 2 months before diagnosis - abdominal pain for at least 4 days per month associated with one/more of the change in evacuation frequency, change in the shape/appearance of stools, if constipation is noticed pain does not resolve with the resolution of constipation - in the absence of organic disease).

SECONDARY OUTCOMES:
Diagnostic accuracy of the patch test with peach juice | At baseline
  The atopy patch test is evaluated through visual inspection 48 hours after patch removal, with an optional second reading at 72 hours to detect delayed reactions.
  The reaction at the application site is assessed based on its intensity and classified according to a semi-quantitative scale:
  - +: erythema with infiltration
  * ++: erythema with a few papules
  * +++: erythema with numerous or widespread papules
  * ++++: erythema with vesicles.
Evaluation of the potential immunomodulatory effect of Chelanik® on blood mononuclear cells: characterization and activation of CD4+ and CD8+ T populations | At baseline
  Flow cytometric analysis
  For the analysis of phenotypes by multiparametric flow cytometry, the following will be used:
  Antibody panels:
  * T cell panel: anti-CD3, anti-CD4, anti-CD8, anti-HLA-DR (anti-CD4, anti-CD8, anti-HLA-DR (anti-CD4, anti-CD8, anti-HLA-DR (anti-CD4, anti-CD4, anti-CD4, anti-CD4, anti-CD4, anti-CD8, anti-HLA-DR (anti T lymphocytes), CD45RA (na.ve lymphocytes), CCR7 (memory T cells) and CD38 (activation).
  * Th1/Th2/Th17 panel: CD3, CD4, CD8, HLA-DR, CCR4 (Th2-associated marker), CCR6 (Th17), CXCR3 (Th1), and CD38 (activation).
  * Regulatory T cell panel: CD3, CD4, CCR4 (Treg migration), CD25 (activation) and CD127.
Evaluation of the potential immunomodulatory effect of Chelanik® on blood mononuclear cells: cytokines production | At baseline
  Cytokine assay by ELISA test Analysis of cytokine expression levels (IL-2, IL-5, IL-13, IL-4, IL-22, IFN-γ, IL-17, TNF-α, IL-10) will be. performed on both serum and supernatants of PBMCs cultures. The concentrations of the individual cytokines will be quantified by ELISA enzyme immunoassay, according to the protocols and recommendations provided by the manufacturer of the kit used.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Traslational Medical Science - University of Naples Federico II, Naples, Italy